CLINICAL TRIAL: NCT02022241
Title: Repeated Injection of GnRH Agonist for Triggering Final Oocyte Maturation in Patients at High Risk of Ovarian Hyperstimulation Syndrome in GnRH Antagonist Protocol
Brief Title: Repeated Injection of GnRH Agonist to Reduce Ovarian Hyperstimulation Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chenshiling (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Comprehensive Strategic Cooperation Project of Guangdong Province and Chinese Academy of Science (Other); Guangzhou Science and Technology Program key projects (Other); National Key Basic Research Development Plan of China (Unknown)
Responsible Party: Sponsor-Investigator, Chenshiling, Professor, M.D., Ph.D., Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Repeated GnRHa trigger
Record Dates: First submitted 2013-12-15; First posted 2013-12-27 (Estimated); Last update posted 2013-12-27 (Estimated); Status verified 2013-12

CONDITIONS: Infertility and at High Risk of OHSS
Keywords: Ovarian Hyperstimulation Syndrome; Luteinizing Hormone; Polycystic Ovarian Syndrome; Ovarian Yield; Ovarian Maturity
MeSH Terms: conditions — Infertility; Ovarian Hyperstimulation Syndrome; Polycystic Ovary Syndrome | interventions — Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Repeated GnRHa (Experimental): Patients were triggered with repeated GnRHa
  Interventions: Drug: triptorelin

INTERVENTIONS:
Drug: triptorelin — 0.2 mg, ih, at night and 0.2 mg, ih, 12 hours later when at least one of the following criteria was reached: (i) serum E2 ≥3500 pg/ml, (ii) ≥18 follicles measuring ≥11 mm.
  Other Names: Diphereline

SUMMARY:
Gonadotropin releasing hormone (GnRH) agonist is sufficient for triggering final oocyte maturation in GnRH antagonist protocol and can significantly reduce incidence of ovarian hyperstimulation syndrome (OHSS) in high-risk patients.

However, lower oocyte yield was reported in patients with lower luteinizing hormone (LH) level post trigger with single injection of GnRH agonist, which might be related to the shorter duration and lower amount of LH induced by GnRH agonist.

Our aim is to study repeated injection of GnRH agonist for preventing OHSS and maintaining clinical outcome in high risk patients who receive controlled ovarian stimulation in GnRH antagonist protocol.

DETAILED DESCRIPTION:
This was a prospective cohort study of all women attending the Center for Reproductive Medicine, Department of Gynecology and Obstetrics, Nanfang Hospital, affiliated with Southern Medical University for in vitro fertilization and/or intracytoplasmic sperm injection . Women at high risk of OHSS who received IVF and/or intracytoplasmic sperm injection (ICSI) treatment with a flexible GnRH antagonist protocol were recruited to participate in this study.

All patients underwent standard ovarian stimulation protocol with gonadotropins, standard individualized adjustment of medication dose, and standard egg retrieval procedure. Patients were triggered with a single bolus of 0.2 mg triptorelin at night and had second injection of 0.2 mg triptorelin 12 hours later when the criteria for administration of the ovulation trigger were met.

ELIGIBILITY:
Inclusion Criteria:

* patients with polycystic ovarian syndrome
* patients with polycystic ovarian morphology on ultrasound
* patients who previously experienced an ovarian stimulation cycle, with a high response to gonadotrophins

Exclusion Criteria:

* patients undergoing coasting
* patients with past ovarian surgery

Max Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate per transfer cycle | 1month post embryo transfer
numbers of patients having OHSS | 2 weeks post trigger with repeated GnRHa
oocyte yield | oocyte retrieval day (34 to 38 hours post the first trigger with GnRHa)
  Oocyte yield was defined as the ratio of the total number of collected oocytes to the number of follicles measuring ≥10 mm on the day of oocyte retrieval.
Oocyte maturity | 24 hours post oocyte retrieval day
  Oocyte maturity was defined as the ratio of metaphase II (MII) oocytes to the number of collected oocytes in the patients undergoing with ICSI.

SECONDARY OUTCOMES:
serum luteinizing hormone level 12 hours post first trigger | 12 hours post trigger with the first injection of GnRHa
serum luteinizing hormone level 24 hours post first trigger | 24 hours post the first injection of GnRHa
fertilization rate | 48 hours post IVF/ICSI
  Fertilization rate was defined as the ratio of normal fertilized oocytes (2PNs) to the number of oocytes used for fertilization (i.e. the denominator in IVF in calculating fertilization rate is all oocytes recovered, but in ICSI it is calculated using only the number of MII oocytes).
implantation rate | 1 month post embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ling Chen, M.D., Ph.D., Study Chair — Nanfang Hospital, Southern Medical University; Xin Chen, M.D., Ph.D., Study Director — Nanfang Hospital, Southern Medical University
Locations (1):
- Center for Reproductive Medicine, Department of Gynecology and Obstetrics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China